CLINICAL TRIAL: NCT03137368
Title: A Randomized Controlled Study to Evaluate Exemestane Tablets Combined With Ovarian Function Suppression/Ablation in Treatment of Premenopausal Breast Cancer Patients With CYP2D6*10 Mutations （STEP）
Brief Title: A Study to Evaluate Exemestane Tablets Combined With Ovarian Function Suppression/Ablation in Treatment of Premenopausal Breast Cancer Patients With CYP2D6*10 Mutations （STEP）
Acronym: STEP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ma Fei, Deputy Director of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-059
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: CYP2D6 Polymorphism
Keywords: ovarian function suppression/ablation; breast cancer; Exemestane; Tamoxifen; CYP2D6*10 mutations
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Tamoxifen

STUDY DESIGN:
Intervention Model Description: randomized, open-label, parallel, active-controlled superiority clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- treatment group (Experimental): Exemestane Tablets combined with ovarian function suppression/ablation
  Interventions: Drug: Exemestane Tablets; Other: ovarian function suppression/ablation; Genetic: CYP2D6*10 gene test
- control group (Active Comparator): Tamoxifen Tablets combined with ovarian function suppression/ablation
  Interventions: Other: ovarian function suppression/ablation; Genetic: CYP2D6*10 gene test; Drug: Tamoxifen

INTERVENTIONS:
Drug: Exemestane Tablets — drug therapy
  Arms: treatment group
Other: ovarian function suppression/ablation — Gonadotropin-releasing hormone analogue Goserelin Injection 3.6mg or Leuprorelin Injection 3.75 mg, a subcutaneous injection should be done every 28±2 days; or Bilateral ovariectomy.
Genetic: CYP2D6*10 gene test — CYP2D6*10 gene test
Drug: Tamoxifen — drug therapy
  Arms: control group

SUMMARY:
This is a multicenter, randomized, open-label, parallel, active-controlled superiority clinical study conducted in early premenopausal estrogen-receptor positive breast cancer patients with CYP2D6*10 mutations. The efficacy and safety of Exemestane Tablets combined with ovarian function suppression/ablation and Tamoxifen Tablets combined with ovarian function suppression/ablation in the treatment of early premenopausal estrogen-receptor positive breast cancer patients with CYP2D6*10 mutations are compared.

DETAILED DESCRIPTION:
The target population for this study is early stage premenopausal estrogen-receptor positive breast cancer patients with CYP2D6*10 mutations. All the potential subjects must provide the informed consent. The subjects who provide the informed consent form (ICF) will enter the screening period, and will be evaluated for the eligibility.

This study expects to enroll 300 subjects, eligible subjects will be randomized at a ratio of 1:1 into treatment group (Exemestane Tablets combined with ovarian function suppression/ablation) or control group (Tamoxifen Tablets combined with ovarian function suppression/ablation).

The subjects who are assigned to treatment group will receive Exemestane Tablet combined with ovarian function suppression/ablation, Exemestane Tablets orally, once a day, one tablet each time (25 mg) and to be taken within 8 weeks from receiving ovarian function suppression treatment or after bilateral ovariectomy, and continue for 5 years or until endpoint event occurs. If the patients are not treated for 5 years because of adverse events (AE) or other reasons, the patient should be followed up until 5 years.

The subjects who are assigned to the control group will receive Tamoxifen Tablets combined with ovarian function suppression/ablation, Tamoxifen Tablets orally, twice a day, one tablet each time (10mg) and to be taken within 8 weeks from receiving ovarian function suppression treatment or after bilateral ovariectomy, and continue for 5 years or until endpoint event occurs. If the patients are not treated for 5 years because of adverse events (AE) or other reasons, the patient should be followed up until 5 years.

The treatment regimen of ovarian function suppression/ablation is as follows: Gonadotropin-releasing hormone analogue Goserelin Injection 3.6mg or Leuprorelin Injection 3.75 mg, a subcutaneous injection will be done every 28±2 days, or bilateral ovariectomy.

According to clinical practice of adjuvant endocrine therapy for Chinese patients with breast cancer, safety and effectiveness of all patients will be evaluated once every 3 months within 2 years after receiving the study treatment, every 6 months in 3 and 4 years, every 12 months in 5 years and 30 days after treatment discontinuation. After randomization, all patients should be regularly checked for signs, symptoms, and evidence of disease recurrence by collecting their medical history, physical examination, and local examination of the breast (specialized physical examination and/or imaging examination). Patients are advised to take a bone mineral density test once a year within five years from 6 months after randomization, and receive calcium or phosphate correspondingly based on the condition. Throughout the study, the adverse events need to be closely monitored, and the frequency and severity of adverse events are recorded as well.

The study results will be statistically analyzed after the study to compare the efficacy and safety variables between the two groups, thus, the superiority of Exemestane Tablets combined with ovarian function suppression/ablation to Tamoxifen Tablets combined with ovarian function suppression/ablation in disease-free survival (DFS) will be demonstrated. Stratified analyses according to lymph-node status and age.

ELIGIBILITY:
Inclusion Criteria:

* Providing informed consent forms voluntarily before screening evaluation;
* For Chinese premenopausal women, her estradiol level must be within the premenopausal level, or the patient meet the following 4 criteria in the prior 6 months: No chemotherapy, Regular menstruation, No use of hormonal, contraceptives, No use of hormone for treatment or for temporary amenorrhea caused by chemotherapy, the estradiol level tested within 8 months after the last dose of chemotherapeutics is within the premenopausal level;
* Patients with invasive breast cancer which has been confirmed by histological examination;
* Complete removal of tumor by surgery without local residual;
* Neoadjuvant chemotherapy before surgery is permitted if the surgery for primary breast cancer is performed within 12 weeks without any further adjuvant chemotherapy, or adjuvant chemotherapy is completed within 8 months;
* Estrogen receptor (ER) and/or progesterone receptor (PR) positive: If the patient has more than one breast tumor lesions, each tumor lesion should be ER and/or PR positive.
* Her-2 negative;
* Genotyping test performed by the central laboratory designated by sponsor with the results confirmed as CYP2D6*10T/T gene mutation.
* Women of childbearing age with negative serum pregnancy test result, and agreeing to adopt highly efficient non-hormonal contraception measure throughout the study;
* Subject without major organ dysfunction, and with normal heart, liver, kidney, lung and other major organ function.

Exclusion Criteria:

* Inflammatory breast cancer;
* Breast cancer patients with supraclavicular lymph nodes metastasis;
* Patients with enlarged internal mammary lymph nodes (except for patients with negative pathologic findings);
* Ovariectomy which is not specified in the study;
* Patients with ovary protection during the chemotherapy;
* Concomitant use of other aromatase inhibitors (not Exemestane);
* Received major surgery which was unrelated to breast cancer within four weeks before randomization, or the patients had not yet fully recovered from such surgery;
* Pregnant or lactating women;
* Known active hepatitis B or hepatitis C or HIV;
* Having difficulty in swallowing oral preparations and gastrointestinal dysfunction;
* Recently had severe and uncontrolled systemic diseases (e.g.: cardiovascular disease, lung disease, or metabolic disease, venous thrombosis with clinical significance);
* Currently or previously suffering from other malignant tumors (except for skin basal cell carcinoma or squamous cell carcinoma, carcinoma in situ of cervix which had been fully treated), unless a radical treatment had been done with the evidence of no-recurrence or metastasis in nearly five years;
* Allergic to any study drug or any ingredients of drug;
* Patient with poor compliance or other conditions which makes the patient unsuitable to participate in this study judged by the investigator.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | the first breast cancer local/distant recurrence, the new breast cancer of the contralateral breast, second primary cancer and the death caused by any reason in 5 years
  It is defined as the time from randomization to the first breast cancer local/distant recurrence, the new breast cancer of the contralateral breast, second primary cancer and the death caused by any reason

SECONDARY OUTCOMES:
Recurrence rate (local or distant) | It will be conducted once every 3 months in the first 2 years during the treatment period, every 6 months in 3 and 4 years, every 12 months in 5 years
  Recurrence rate (local or distant) is defined as breast cancer local or distant recurrence rate in patients from two groups
Overall survival (OS) | It will be conducted once every 3 months in the first 2 years during the treatment period, every 6 months in 3 and 4 years, every 12 months in 5 years
  OS is defined as the time from randomization to death due to any reasons
Incidence of Treatment-Emergent Adverse Events | It will be conducted once every 3 months in the first 2 years during the treatment period, every 6 months in 3 and 4 years, every 12 months in 5 years
  Results of AE/serious adverse event (SAE), clinical lab tests, 12 lead ECG, vital signs and physical examination will be evaluated throughout the study to monitor the safety of subjects

OTHER OUTCOMES:
Breast cancer free survival | It will be conducted once every 3 months in the first 2 years during the treatment period, every 6 months in 3 and 4 years, every 12 months in 5 years
  Breast cancer free survival is defined as the time from randomization to the first observation of breast cancer local/distant recurrence or occurrence of contralateral breast cancer
Distant relapse free survival | It will be conducted once every 3 months in the first 2 years during the treatment period, every 6 months in 3 and 4 years, every 12 months in 5 years
  Distant relapse free survival is defined as the time from randomization to the first observation of breast cancer distant recurrence
The occurrence rate of the contralateral breast cancer | It will be conducted once every 3 months in the first 2 years during the treatment period, every 6 months in 3 and 4 years, every 12 months in 5 years
  The occurrence rate of the contralateral breast cancer is defined as contralateral breast cancer occurrence rate in patients from two groups after randomization
the psychosocial factors in patients with breast cancer | It will be conducted once every 3 months in the first 2 years during the treatment period, every 6 months in 3 and 4 years, every 12 months in 5 years
  To investigate the psychosocial changes in patients with breast cancer during endocrine therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CancerIHCAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schroth W, Goetz MP, Hamann U, Fasching PA, Schmidt M, Winter S, Fritz P, Simon W, Suman VJ, Ames MM, Safgren SL, Kuffel MJ, Ulmer HU, Bolander J, Strick R, Beckmann MW, Koelbl H, Weinshilboum RM, Ingle JN, Eichelbaum M, Schwab M, Brauch H. Association between CYP2D6 polymorphisms and outcomes among women with early stage breast cancer treated with tamoxifen. JAMA. 2009 Oct 7;302(13):1429-36. doi: 10.1001/jama.2009.1420. PMID 19809024
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Result] Williams C, Brunskill S, Altman D, Briggs A, Campbell H, Clarke M, Glanville J, Gray A, Harris A, Johnston K, Lodge M. Cost-effectiveness of using prognostic information to select women with breast cancer for adjuvant systemic therapy. Health Technol Assess. 2006 Sep;10(34):iii-iv, ix-xi, 1-204. doi: 10.3310/hta10340. PMID 16959170
- [Result] Gansler T, Ganz PA, Grant M, Greene FL, Johnstone P, Mahoney M, Newman LA, Oh WK, Thomas CR Jr, Thun MJ, Vickers AJ, Wender RC, Brawley OW. Sixty years of CA: a cancer journal for clinicians. CA Cancer J Clin. 2010 Nov-Dec;60(6):345-50. doi: 10.3322/caac.20088. PMID 21075954
- [Result] Buzdar A. The place of chemotherapy in the treatment of early breast cancer. Br J Cancer. 1998 Sep;78 Suppl 4(Suppl 4):16-20. doi: 10.1038/bjc.1998.757. PMID 9741784
- [Result] Dezentje VO, Guchelaar HJ, Nortier JW, van de Velde CJ, Gelderblom H. Clinical implications of CYP2D6 genotyping in tamoxifen treatment for breast cancer. Clin Cancer Res. 2009 Jan 1;15(1):15-21. doi: 10.1158/1078-0432.CCR-08-2006. PMID 19118028
- [Result] Blackburn HL, Ellsworth DL, Shriver CD, Ellsworth RE. Role of cytochrome P450 genes in breast cancer etiology and treatment: effects on estrogen biosynthesis, metabolism, and response to endocrine therapy. Cancer Causes Control. 2015 Mar;26(3):319-32. doi: 10.1007/s10552-014-0519-7. Epub 2015 Jan 3. PMID 25554091
- [Result] Brauch H, Schroth W, Eichelbaum M, Schwab M, Harbeck N; in cooperation with the AGO TRAFO Comission. Clinical Relevance of CYP2D6 Genetics for Tamoxifen Response in Breast Cancer. Breast Care (Basel). 2008;3(1):43-50. doi: 10.1159/000114642. Epub 2008 Feb 22. PMID 20824020
- [Result] Jin Y, Desta Z, Stearns V, Ward B, Ho H, Lee KH, Skaar T, Storniolo AM, Li L, Araba A, Blanchard R, Nguyen A, Ullmer L, Hayden J, Lemler S, Weinshilboum RM, Rae JM, Hayes DF, Flockhart DA. CYP2D6 genotype, antidepressant use, and tamoxifen metabolism during adjuvant breast cancer treatment. J Natl Cancer Inst. 2005 Jan 5;97(1):30-9. doi: 10.1093/jnci/dji005. PMID 15632378
- [Result] Goetz MP, Rae JM, Suman VJ, Safgren SL, Ames MM, Visscher DW, Reynolds C, Couch FJ, Lingle WL, Flockhart DA, Desta Z, Perez EA, Ingle JN. Pharmacogenetics of tamoxifen biotransformation is associated with clinical outcomes of efficacy and hot flashes. J Clin Oncol. 2005 Dec 20;23(36):9312-8. doi: 10.1200/JCO.2005.03.3266. PMID 16361630
- [Result] Schroth W, Antoniadou L, Fritz P, Schwab M, Muerdter T, Zanger UM, Simon W, Eichelbaum M, Brauch H. Breast cancer treatment outcome with adjuvant tamoxifen relative to patient CYP2D6 and CYP2C19 genotypes. J Clin Oncol. 2007 Nov 20;25(33):5187-93. doi: 10.1200/JCO.2007.12.2705. PMID 18024866
- [Result] Thompson AM, Johnson A, Quinlan P, Hillman G, Fontecha M, Bray SE, Purdie CA, Jordan LB, Ferraldeschi R, Latif A, Hadfield KD, Clarke RB, Ashcroft L, Evans DG, Howell A, Nikoloff M, Lawrence J, Newman WG. Comprehensive CYP2D6 genotype and adherence affect outcome in breast cancer patients treated with tamoxifen monotherapy. Breast Cancer Res Treat. 2011 Jan;125(1):279-87. doi: 10.1007/s10549-010-1139-x. Epub 2010 Sep 1. PMID 20809362
- [Result] Margolin S, Lindh JD, Thoren L, Xie H, Koukel L, Dahl ML, Eliasson E. CYP2D6 and adjuvant tamoxifen: possible differences of outcome in pre- and post-menopausal patients. Pharmacogenomics. 2013 Apr;14(6):613-22. doi: 10.2217/pgs.13.47. PMID 23570465
- [Result] Bradford LD. CYP2D6 allele frequency in European Caucasians, Asians, Africans and their descendants. Pharmacogenomics. 2002 Mar;3(2):229-43. doi: 10.1517/14622416.3.2.229. PMID 11972444
- [Result] Sistonen J, Sajantila A, Lao O, Corander J, Barbujani G, Fuselli S. CYP2D6 worldwide genetic variation shows high frequency of altered activity variants and no continental structure. Pharmacogenet Genomics. 2007 Feb;17(2):93-101. doi: 10.1097/01.fpc.0000239974.69464.f2. PMID 17301689
- [Result] Qian JC, Xu XM, Hu GX, Dai DP, Xu RA, Hu LM, Li FH, Zhang XH, Yang JF, Cai JP. Genetic variations of human CYP2D6 in the Chinese Han population. Pharmacogenomics. 2013 Nov;14(14):1731-43. doi: 10.2217/pgs.13.160. PMID 24192122
- [Result] Xu Y, Sun Y, Yao L, Shi L, Wu Y, Ouyang T, Li J, Wang T, Fan Z, Fan T, Lin B, He L, Li P, Xie Y. Association between CYP2D6 *10 genotype and survival of breast cancer patients receiving tamoxifen treatment. Ann Oncol. 2008 Aug;19(8):1423-1429. doi: 10.1093/annonc/mdn155. Epub 2008 Apr 11. PMID 18407954
- [Result] Francis PA, Regan MM, Fleming GF, Lang I, Ciruelos E, Bellet M, Bonnefoi HR, Climent MA, Da Prada GA, Burstein HJ, Martino S, Davidson NE, Geyer CE Jr, Walley BA, Coleman R, Kerbrat P, Buchholz S, Ingle JN, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Colleoni M, Viale G, Coates AS, Goldhirsch A, Gelber RD; SOFT Investigators; International Breast Cancer Study Group. Adjuvant ovarian suppression in premenopausal breast cancer. N Engl J Med. 2015 Jan 29;372(5):436-46. doi: 10.1056/NEJMoa1412379. Epub 2014 Dec 11. PMID 25495490
- [Result] Pagani O, Regan MM, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Perez EA, Ciruelos E, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Pinotti G, Puglisi F, Crivellari D, Ruhstaller T, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Bernhard J, Luo W, Ribi K, Viale G, Coates AS, Gelber RD, Goldhirsch A, Francis PA; TEXT and SOFT Investigators; International Breast Cancer Study Group. Adjuvant exemestane with ovarian suppression in premenopausal breast cancer. N Engl J Med. 2014 Jul 10;371(2):107-18. doi: 10.1056/NEJMoa1404037. Epub 2014 Jun 1. PMID 24881463
- [Result] Janni W, Hepp P. Adjuvant aromatase inhibitor therapy: outcomes and safety. Cancer Treat Rev. 2010 May;36(3):249-61. doi: 10.1016/j.ctrv.2009.12.010. Epub 2010 Feb 4. PMID 20133065